CLINICAL TRIAL: NCT03718026
Title: The Reliability, Validity, and Responsiveness of the Timed 360° Turn Test Test in Patients With Multiple Sclerosis
Brief Title: The Reliability, Validity, and Responsiveness of the Timed 360° Turn Test in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fatih Söke, Research Assistant, Gazi University
Other Study IDs: 438
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: The timed 360° turn test; Multiple sclerosis; reliability; validity
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Patients with Multiple Sclerosis: * The timed 360° turn test
  * Berg Balance Scale
  * Timed Up and Go test
  * Functional Reach Test
  * One-leg stance test
  * Four square step test
  Interventions: Other: The timed 360° turn test
- Healthy Controls: -The timed 360° turn test
  Interventions: Other: The timed 360° turn test

INTERVENTIONS:
Other: The timed 360° turn test — * The timed 360° turn test: Each participant turns around in place in a standing position for both sides.
  * Berg Balance Scale: It has 14 items, each of which is scored from 0 (i.e, severely impaired balance) to 4 (i.e., no balance impairment).
  * Timed Up and Go test: It requires individual to stand up from an armed chair, walk 3m, turn around, walk back to the armed chair, and sit down again.
  * Functional Reach Test: It measures the maximum distance an individual is able to reach forward beyond arm's length in the standing position when maintaining a fixed base of support.
  * One-leg stance test: Individuals were asked to stand on either their left or right leg.
  * Four square step test: It requires an individual to step over obstacles in various directions including forward, backward, and sideways.
  Other Names: Berg Balance Scale, Timed Up and Go test, Functional Reach Test, One-leg stance test, Four square step test

SUMMARY:
The aim of the study is to investigate reliability, validity, and responsiveness of the timed 360° turn test in patients with Multiple Sclerosis.

DETAILED DESCRIPTION:
At baseline, the timed 360° turn test, Berg Balance Scale, Timed Up and Go test, Functional Reach Test, Four Square Step Test, and One-legged Stance Test is applied to the Multiple Sclerosis group. The timed 360° turn test is repeated after seven days from the first application in patients with Multiple Sclerosis. Healthy controls are going to perform only the timed 360° turn test.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years,
* neurologist-diagnosed Multiple Sclerosis,
* Expanded Disability Status Scale (EDSS) score < 7,
* able to walk 20 m with or without aids,
* no MS exacerbation within the last 2 months,
* use of stable medication in the last 2 months.

Exclusion Criteria:

* other neurologic disorder,
* Pregnancy,
* orhopedic problems affecting gait and stance,
* visual, auditory, orientational problems that could affect study results,
* Cardiovascular, pulmonary, and humoral disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Sclerosis who apply to Gazi University, Department of Physiotherapy and Rehabilitation will be invited to this study.
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
The timed 360° turn test | 1 minute
  The timed 360° turn test evaluates turning ability. Higher durations indicate worse turning performance.

SECONDARY OUTCOMES:
Berg Balance Scale | 10 minutes
  Berg Balance Scale assesses functional balance. It consists of 14 functional tasks rated on a 5-point scale ranging from 0 to 4. The maximum score is 56 points. Higher scores indicate better functional balance.
Timed Up and Go test | 1 minute
  Timed Up and Go test evaluates functional mobility. Higher durations indicate worse functional mobility.
Functional Reach Test | 1 minute
  Functional Reach Test is used to evaluate limits of stability. Higher distances indicate better limits of stability.
Four Square Step Test | 1 minute
  Four Square Step Test is used to assess dynamic balance. Higher durations indicate worse dynamic balance.
One Leg Stance Test | 3 minutes
  One Leg Stance Test evaluates postural stability. Higher durations indicate better postural stability.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Söke, Principal Investigator — Gazi University
Locations (1):
- Fatih Söke, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adusumilli G, Lancia S, Levasseur VA, Amblee V, Orchard M, Wagner JM, Naismith RT. Turning is an important marker of balance confidence and walking limitation in persons with multiple sclerosis. PLoS One. 2018 Jun 7;13(6):e0198178. doi: 10.1371/journal.pone.0198178. eCollection 2018. PMID 29879144
- [Background] Spain RI, St George RJ, Salarian A, Mancini M, Wagner JM, Horak FB, Bourdette D. Body-worn motion sensors detect balance and gait deficits in people with multiple sclerosis who have normal walking speed. Gait Posture. 2012 Apr;35(4):573-8. doi: 10.1016/j.gaitpost.2011.11.026. Epub 2012 Jan 25. PMID 22277368
- [Background] Gunn H, Creanor S, Haas B, Marsden J, Freeman J. Frequency, characteristics, and consequences of falls in multiple sclerosis: findings from a cohort study. Arch Phys Med Rehabil. 2014 Mar;95(3):538-45. doi: 10.1016/j.apmr.2013.08.244. Epub 2013 Sep 18. PMID 24055784
- [Background] Cameron MH, Asano M, Bourdette D, Finlayson ML. People with multiple sclerosis use many fall prevention strategies but still fall frequently. Arch Phys Med Rehabil. 2013 Aug;94(8):1562-6. doi: 10.1016/j.apmr.2013.01.021. Epub 2013 Feb 4. PMID 23391522